CLINICAL TRIAL: NCT01548885
Title: Evaluation of Blood Glucose Meter Systems - NACT Study
Brief Title: Comparison Evaluation of Blood Glucose Meter Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-PRO-2012-001-01
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Staff Test BGMSs (Experimental): All testing and lancings were performed by the study staff; subjects did not perform any lancing or self-testing in this study. Study Staff lanced the fingers of subjects and tested the blood samples using five Blood Glucose Monitoring Systems(BGMS): FreeStyle Freedom Lite® BGMS; ACCU-CHEK® Aviva BGMS; TRUEtrack® BGMS; OneTouch® Ultra®2 BGMS; CONTOUR® NEXT EZ BGMS.
  Interventions: Device: CONTOUR® NEXT EZ BGMS; Device: FreeStyle Freedom Lite® BGMS; Device: ACCU-CHEK® Aviva BGMS; Device: TRUEtrack® BGMS; Device: OneTouch® Ultra®2 BGMS

INTERVENTIONS:
Device: CONTOUR® NEXT EZ BGMS — Study staff performed Blood Glucose (BG) testing with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). Performance of CONTOUR® NEXT EZ BGMS was evaluated across the glucose range of the BGMs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: FreeStyle Freedom Lite® BGMS — Study staff performed Blood Glucose (BG) testing with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). Performance of FreeStyle Freedom Lite® BGMS was evaluated across the glucose range of the BGMs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: ACCU-CHEK® Aviva BGMS — Study staff performed Blood Glucose (BG) testing with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). Performance of ACCU-CHEK® Aviva BGMS was evaluated across the glucose range of the BGMs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: TRUEtrack® BGMS — Study staff performed Blood Glucose (BG) testing with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). Performance of TRUEtrack® BGMS was evaluated across the glucose range of the BGMs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: OneTouch® Ultra®2 BGMS — Study staff performed Blood Glucose (BG) testing with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). Performance of OneTouch® Ultra®2 BGMS was evaluated across the glucose range of the BGMs. All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

SUMMARY:
The purpose of this study was to evaluate the performance of one investigational Bayer Blood Glucose meter (with investigational Bayer test strips) and four Blood Glucose Monitoring Systems from other companies. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer). Performance of the five systems was evaluated across the glucose range of the BGMSs using capillary blood. All testing and lancing were performed by study staff and some blood samples were glycolyzed to lower the glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 years of age or older
* Willing to complete all study procedures

Exclusion Criteria:

* Blood Borne infections like hepatitis or HIV or infections such as tuberculosis
* Hemophilia or any other bleeding disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Staff Test BGMSs: All testing and lancings were performed by the study staff; subjects did not perform any lancing or self-testing in this study. Study Staff lanced the fingers of subjects and tested the blood samples using five Blood Glucose Monitoring Systems(BGMS): FreeStyle Freedom Lite® BGMS; TRUEtrack® BGMS; OneTouch® Ultra®2 BGMS; ACCU-CHEK® Aviva BGMS; CONTOUR® NEXT EZ BGMS.
Period: Overall Study
Arm/Group | Study Staff Test BGMSs
Started | 146
Completed | 146
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Per protocol
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 146
Age, Continuous [Median (Full Range); unit: years] | 62 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 61
Region of Enrollment [Number; unit: participants]
  United States | 146

OUTCOME MEASURES:

1. Primary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) Across the Overall Tested Glucose Range
Description: Using the overall Blood Glucose(BG) range (24 to 386mg/dL), the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI laboratory reference values were compared. MARD is calculated from the sum of all |(BG meter)-(BG reference)| / (BG Reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all five BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD value indicates smaller difference between meter value and the reference value . Higher MARD value indicates larger difference between meter value and the reference value.
Time Frame: 10 hours
Population: Same number 388(393-3-2)BG results possible for each BGMS.Subjects provided 1,2,or 3 capillary samples-total 393 samples. 3 glycolyzed samples were not analyzed - glycolysis exceeded the protocol-defined time. All meter data for 2 glycolyzed samples were not evaluable (not analyzed)- their YSI results were less than the meter operating ranges.
Measure: Mean (95% Confidence Interval); unit: percentage
Units Other Than Participants: BG test results
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 146
Number analyzed (BG test results) | 388
percentage
  CONTOUR® NEXT EZ BGMS | 4.7 [0 to 11.4]
  ACCU-CHEK® Aviva BGMS | 6.3 [0 to 13.0]
  FreeStyle Freedom Lite® BGMS | 18.3 [11.6 to 25.0]
  OneTouch® Ultra®2 BGMS | 23.4 [16.7 to 30.1]
  TRUEtrack® BGMS | 26.2 [19.5 to 32.9]

2. Secondary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) Across the Low Glucose Range (<70mg/dL)
Description: Using fresh and glycolyzed samples with Blood Glucose(BG) below 70 mg/dL, the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI laboratory reference values were compared. MARD is calculated from the sum of all |(BG meter)-(BG reference)| / (BG Reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all five BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD value indicates smaller difference between meter value and the reference value . Higher MARD value indicates larger difference between meter value and the reference value.
Time Frame: 10 hours
Population: Same number (190) of BG results was possible for each BGMS. Subjects provided 1,2,or 3 capillary samples, of which 190 samples were less than 70 mg/dL.
Measure: Mean (95% Confidence Interval); unit: percentage
Units Other Than Participants: BG test results
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 146
Number analyzed (BG test results) | 190
percentage
  CONTOUR® NEXT EZ BGMS | 0.7 [0 to 6.8]
  ACCU-CHEK® Aviva BGMS | 2.5 [0 to 8.7]
  FreeStyle Freedom Lite® BGMS | 18.3 [12.1 to 28.6]
  OneTouch® Ultra®2 BGMS | 22.4 [16.2 to 28.6]
  TRUEtrack® BGMS | 33.2 [27.1 to 39.4]

ADVERSE EVENTS:
Arm/Group | Study Staff Test BGMSs
Serious Adverse Events (participants affected / at risk) | 0/146
Other Adverse Events (participants affected / at risk) | 4/146
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Staff Test BGMSs (N=146)
hypoglycemia (Endocrine disorders) | 4 (4) — Mild, Not device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes